CLINICAL TRIAL: NCT01168726
Title: Protective Behavioral Strategies and Brief Alcohol Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Matthew P. Martens, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protective Behaviors; 1R21AA016779-01A2 (NIH)
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protective Behavioral Strategies (Experimental): Personalized feedback on use of protective behavioral strategies.
  Interventions: Behavioral: Protective Behavioral Strategies
- Personalized Normative Feedback (Experimental): Personalized feedback on how one's own drinking compares to relevant norms.
  Interventions: Behavioral: Personalized Normative Feedback
- Alcohol Education (Active Comparator): Educational information about harms associated with heavy drinking.
  Interventions: Behavioral: Alcohol Education

INTERVENTIONS:
Behavioral: Protective Behavioral Strategies — Personalized feedback on use of protective behavioral strategies.
  Arms: Protective Behavioral Strategies
Behavioral: Personalized Normative Feedback — Personalized feedback on how one's own drinking compares to relevant norms.
  Arms: Personalized Normative Feedback
Behavioral: Alcohol Education — Educational information about harms associated with heavy drinking.
  Arms: Alcohol Education

SUMMARY:
Excessive college student drinking represents an important public health problem for both the students themselves and those with whom they interact. The objective of this research is to better understand how to reduce such high-risk drinking by improving prevention and treatment programs, which will provide an overall public health benefit. Subjects in the study will be randomized to one of two brief intervention conditions or an education-only control condition. It is hypothesized that those in the intervention conditions will report greater reductions in alcohol use and alcohol-related problems than those in the control condition.

DETAILED DESCRIPTION:
The primary objective of this project is to examine factors that are associated with the effectiveness of intervention programs designed to reduce high-risk drinking among heavy drinking college students. Previous research has found similar effect sizes for different types of multi-component, brief interventions among college students, but little research has assessed the degree to which specific components of such interventions are associated with intervention outcomes. One common component of motivational enhancing interventions among college students involves providing cognitive-behavioral self-control strategies designed to reduce one's use of alcohol, which we term "protective behavioral strategies" (PBS). However, there are two important factors that limit our understanding of the effects of PBS on client outcomes. First, the use of these strategies in motivational enhancing programs has generally not been assessed in a systematic manner, due in part to the fact that until recently a standardized measure of such strategies did not exist. Second, researchers have yet to conduct studies that dismantle the specific effects associated with the PBS component on client outcomes. That is, studies have not tested interventions with and without assessment and feedback regarding a client's use of PBS. Participants in this project will be "at-risk" college student drinkers who will be assigned to one of three conditions: a brief intervention that includes a focus on PBS, a brief intervention that does not include this focus, and an education-only control condition. Participant will complete self-report measures of alcohol-related variables at baseline, 30-day, and 6-month follow-ups. Mixed-model analyses will be used to determine the effectiveness of the intervention programs, and structural equation modeling will be used to determine if increases in PBS result in reductions in alcohol use/alcohol-related problems.

ELIGIBILITY:
Inclusion Criteria:

* At least one binge drinking episode in the preceding month

Exclusion Criteria:

* At-risk for alcohol dependence or major depressive disorder

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Martens, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Protective Behavioral Strategies: Protective Behavioral Strategies Feedback: Personalized feedback on use of protective behavioral strategies.
Period: Overall Study
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Started | 111 | 121 | 133
Completed | 103 | 112 | 128
Not Completed | 8 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education | Total
Number analyzed (Participants) | 111 | 121 | 133 | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 121 | 133 | 365
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.95 (1.36) | 20.12 (1.38) | 20.20 (1.31) | 20.10 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 50 | 48 | 127
  Male | 82 | 71 | 85 | 238
Region of Enrollment [Number; unit: participants]
  United States | 111 | 121 | 133 | 365

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Week
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Number analyzed (Participants) | 111 | 121 | 133
drinks per week | 12.55 (8.96) | 9.57 (8.78) | 13.74 (10.77)

2. Primary Outcome: Rutgers Alcohol Problems Index (RAPI)
Description: Total scores on an alcohol problems scale. Possible score range = 0-92. Higher scores are indicative of more alcohol-related problems.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Number analyzed (Participants) | 111 | 121 | 133
units on a scale | 7.68 (7.25) | 7.76 (9.42) | 8.91 (9.17)

3. Secondary Outcome: Drinking Norms Rating Form
Description: Perceived drinking among other students, represented by standardized scores on the Drinking Norms Rating Form. Higher values indicate that the individual perceives higher levels of drinking among other students. Because the scores are standardized their is no hypothetical minimum or maximum, and the scale is standardized with a mean of 0 and standard deviation of 1. So, a mean value of 1.52 means that participants in that condition had an average score that was 1.52 standard deviation above the overall mean of the sample.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale (standardized)
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Number analyzed (Participants) | 111 | 121 | 133
units on a scale (standardized) | 1.52 (3.52) | -2.71 (2.57) | 1.20 (3.79)

4. Secondary Outcome: Protective Behavioral Strategies Scale.
Description: Use of protective behavioral strategies related to alcohol use. Higher scores indicate more use of the strategies. A total score was calculated by summing the three subscale scores on the measure (range = 3-18).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Number analyzed (Participants) | 111 | 121 | 133
units on a scale | 12.41 (1.94) | 12.14 (2.24) | 11.44 (2.01)

ADVERSE EVENTS:
Arm/Group | Protective Behavioral Strategies | Personalized Normative Feedback | Alcohol Education
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/121 | 0/133
Other Adverse Events (participants affected / at risk) | 0/111 | 0/121 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No